CLINICAL TRIAL: NCT06729554
Title: Education & Care in RARE - Efficacy of Targeted Psychoeducational Intervention to Improve Knowledge About Rare Diseases and to Promote Mental Health Among Pediatric Rare Disease Patients
Brief Title: Education & Care in RARE: Efficacy of Targeted Psychoeducational Intervention Among Pediatric Rare Disease Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Julia Vodopiutz, MD ap Prof, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1870/2024 ethics committee Nr; 010270-FGÖ (Other Grant/Funding Number: The Austrian Health Promotion (FGÖ))
Record Dates: First submitted 2024-12-03; First posted 2024-12-11 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Orphan Diseases; Rare Disorders; Pediatric Diseases; Inborn Errors of Metabolism Disorders
Keywords: Rare diseases; ultra-rare diseases; psychoeducation in pediatrics; psychoeducation for alle rare diseases; rare pediatric diseases; orphan diseases psychoeducation; rare disease burden; waiting list control study
MeSH Terms: conditions — Rare Diseases | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: This study is a prospective, multicenter, randomized and controlled study with a waiting list. Intervention is psychoeducation using Education & Care in RARE, a short-term, structured, resource-oriented and child-friendly psychoeducation program for children and adolescents with rare diseases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (IG) (Experimental): Participants are randomized in an intervention group (IG) and a waiting list control group (WLG). The IG receive the intervention with Education & Care in RARE (all children) and complete the identical questionnaires (all children and their legal guardians) immedeately after inclusion.
  Interventions: Other: Education & Care in RARE
- Waiting List Control Group (WLG) (Active Comparator): Compared to the IG, the WLG receives the intervention with Education & Care in RARE with a time delay (8-12 weeks later) and has one additional appointment for questionnaire evaluation before start of the intervention.
  Interventions: Other: Education & Care in RARE

INTERVENTIONS:
Other: Education & Care in RARE — Education & Care in RARE (https://www.youtube.com/watch?v=R3fr-q-6JIw) is a short-term, structured, resource-oriented and child-friendly psychoeducation program for children and adolescents with rare diseases. It promotes knowledge and competence on rare diseases in children in order to reduce the psychosocial rare disease burden and to improve individual self-competence in managing the rare disease and to improve their quality of life. Education & Care in RARE can be used for all pediatric rare diseases. This has the great advantage that users only need to be trained in the use of one program.

SUMMARY:
"Rare Diseases" is an umbrella term including more than 8.000 different diseases which individually affect only a small percentage of people. Rare diseases predominantly affect children and adolescents and are associated with high medical and psychosocial burden of disease.

The investigators invented Education & Care in RARE - a short-term, structured, resource-oriented and child-friendly psychoeducation program for children and adolescents with rare diseases.

This study is a prospective, multicenter, randomized and controlled study with a waiting list. Aim of the study is to investigate the efficacy of Education & Care in RARE on knowledge about rare diseases and on mental health well-being in pediatric rare disease patients, compared to a control group.

In this study participants are randomized in an intervention group and a waiting list control group. Both study groups thus receive the psychoeducation with Education & Care in RARE and complete the identical questionnaires. Compared to the Intervention group, the waiting list control group receives the intervention with a time delay (8-12 weeks later) and has one additional appointment for questionnaire evaluation before start of the psychoeducation.

DETAILED DESCRIPTION:
1. Background 1.1. Rare diseases Rare diseases are defined as serious diseases which affect only a very small number of people compared to the general population. The more than 8.000 different rare diseases most often affect children and encompass an enormous heterogenous clinical spectrum associated mostly with a chronic or progressive disease course. In addition to the clinical and economic burden of a chronic disease, patients with rare diseases faces also the "rare disease burden" which describes associated problems caused by rarity of the disease. 1-3While advances in rare disease research have significantly improved the diagnostic and therapeutic strategies in rare diseases, psychosocial care is still not part of routine care in rare diseases. 4 1.2. Own previous work The investigator team is highly experienced in both, the molecular characterization 5-16 and the clinical care 17-21 of rare and ultra-rare diseases and in psychosocial care 22-27 of pediatric patients in acute and chronic stress situations. Based on this experience the investigators developed a psycho-educational intervention program for children and adolescents affected by a rare disease named "Education & Care in RARE" Figure 1.

   Education & Care in RARE (https://www.youtube.com/watch?v=R3fr-q-6JIw) is a short-term, structured, resource-oriented and child-friendly psychoeducation program for children and adolescents with rare diseases. It promotes knowledge and competence on rare diseases in children in order to reduce the psychosocial rare disease burden and to improve individual self-competence in managing the rare disease and to improve their quality of life. Education & Care in RARE can be used for all pediatric rare diseases. This has the great advantage that users only need to be trained in the use of one program. Figure 1 Education & Care in RARE is used during clinical care at the outpatient clinic for clinical genetics, Department of Pediatrics and Adolescent Medicine, Division of Pediatric Pulmonology, Allergology and Endocrinology. Education & Care in RARE is currently not available in routine care outside of this specialized outpatient clinic. Affected children who have completed Education & Care in RARE during clinical care, have rated this as a very helpful and supportive program. To date, there has been no study on the effectiveness of Education & Care in RARE.
2. Aims and hypotheses of the study 2.1. Aims This study aims to investigate the efficacy of Education & Care in RARE on knowledge about rare diseases and on mental health well-being in pediatric rare disease patients.

   As a primary objective the investigators will evaluate

   > The effect of Education & Care in RARE on participants' self-rating scales regarding knowledge about rare diseases and well-being, compared to a control group.

   As secondary objectives the investigators will evaluate
   * The effect of Education & Care in RARE on expert-rating scales regarding participants' knowledge about rare diseases and competences to cope with rare-disease specific challenges, compared to a control group.
   * The effect of Education & Care in RARE on generic Quality of Life and mental health well-being questionnaires, compared to a control group.
   * Moderating effects (such as age, rare disease diagnosis, additional diagnosis) on the efficacy of Education & Care in RARE
   * The long-term effect of Education & Care in RARE on participants' knowledge about rare diseases and on mental health well-being.
   * Differences in Quality of Life and mental health well-being of children and adolescents with rare disease, compared to norm data.
   * Since this is the first study on Education & Care in RARE, we will also evaluate the satisfaction with the intervention for the intervention groups and for the applying experts.

   2.2. Hypotheses

   Specifically, the investigators will test the following hypotheses:

   Primary hypothesis:

   • H1: Education & Care in RARE will have a different impact on the change in rare disease specific knowledge and well-being (Rare Disease Specific Self-Rating Scale), between the study time points T0 and T1, in the intervention group compared to the waitlist control group.

   Secondary hypotheses:
   * H2: Education & Care in RARE will have a different impact on the change in experts' opinion regarding participant's knowledge and competences (Rare Disease Specific Expert-Rating Scale), between the study time points T0 and T1, in the intervention group compared to the waitlist control group.
   * H3: Education & Care in RARE will have a different impact on the change of Quality of Life (KINDLR self-report) and mental-health well-being (SDQR self-report), between the study time points T0 and T1, in the intervention group compared to the waitlist control group.
   * H4: Participants' age (H4a), educational level (H4b), and intellectual ability (H4c) will moderate the effect of Education & Care in RARE on participants' rare diseases knowledge and well-being (Rare Disease Specific Self-Rating Scale, Rare Disease Specific Expert-Rating Scale). Education & Care in RARE will have stronger effects for older participants, participants with higher educational levels and participants with normal intellectual ability.
   * H5: Education & Care in RARE will have a different impact on the long-term change in knowledge and well-being (Rare Disease Specific Self-Rating Scale, H5a), experts' opinion regarding participant's knowledge and competences (Rare Disease Specific Expert-Rating Scale, H5b) and change of Quality of Life (KINDLR self-report, KINDLR third-party-report, H5c) and mental-health well-being (SDQR self-report, SDQR third-party-report, H5d) , between the study time points T0 and T2 in the intervention group.

   H6: Rare diseases affect Quality of Life (KINDLR self-report, KINDLR third-party-report) and mental-health well-being (SDQR self-report, SDQR third-party-report,) in pediatric rare disease patients, at T0 in the intervention and in the waitlist control group, compared to norm data.
3. Originality and scientific innovation

   During a 6-year period, from 2018-2024 at MUW, based on the expertise of a highly specialized, multiprofessional and multidisciplinary expertise team, the investigators invented Education & Care in RARE:

   https://www.youtube.com/watch?v=R3fr-q-6JIw Education & Care in RARE is the first targeted psychoeducational program which can be applied in all 8.000 rare diseases. This has the great advantage that users only need to be trained in the use of one program.

   Education & Care in RARE is a short-term, structured, resource-oriented and child-friendly psychoeducation program for children and adolescents with rare diseases. It promotes knowledge and competence on rare diseases in children in order to reduce the psychosocial rare disease burden and to improve individual self-competence in managing the rare disease and to improve their quality of life. Education & Care in RARE can be used for all pediatric rare diseases.
4. Research design 4.1. Type of study This study is a prospective 2-arm waitlist randomized controlled trial, that will test the efficacy of a targeted psychoeducation with Education & Care in RARE in pediatric rare diseases patients. Participants will be randomly assigned (1:1 allocation) to either the intervention group, which benefits from the Education & Care in RARE program, or a waiting list control group that will also receive the Education & Care in RARE intervention after the intervention group finishes it. The 2 independent groups (IG versus WLG) will be evaluated at different measurement times (in IG: baseline T0, the postintervention time point T1, and 3-6 month follow-up T2; in WLG baseline T0 and T1, the postintervention time point T2, and 3-6 month follow-up T3).

4.2. Intervention

Intervention in this study is a targeted psychoeducation for pediatric rare diseases using Education & Care in RARE. To enable standardized application of the intervention, the implementation and objectives of the intervention using Education & Care in RARE are defined as followed:

4.2.1. Standardization - application of the intervention

* All participating centers completed a one-day workshop to learn how to use the Education & Care in RARE program.
* The intervention (Education & Care in RARE program) is done in a one-to-one setting (trained member of the medical care team and the pediatric study participant).
* Consultation of participant's medical and psychosocial care team, before applying the intervention, to ensure quality-assured knowledge transfer regarding the specific rare disease of the individual study participant.
* Execution of the Education & Care in RARE program from front to back (Chapter 1-4) according to the Education & Care in RARE Manual
* Completion of Education & Care in RARE within up to 8 weeks. Within this 8-week period a variable number of sessions and a variable duration of the sessions can be used to complete the Education & Care in RARE program.

4.2.2. Standardization - aims of the intervention

Basic learning objectives of the intervention, which should be achieved by the intervention are defined as followed:

* Establishment of 3 names for the rare disease

  * rare disease name within the medical system
  * rare disease name within the patient's social system
  * what to say if the patient does not want to talk about the rare disease
* Acquisition of knowledge on the underlying rare diseases (eg. knowledge about the emergency card, knowledge about special risk factors, knowledge about etiology, etiology of disease symptoms and healthy body functions)
* Acquisition of knowledge on rare diseases in general
* Acquisition of competences in dealing with the rare disease in daily life
* Emotional relief of the child 4.3. Setting This multicenter trial will be performed at pediatric centers in Austria who are specially experienced in diagnostics and therapeutics of pediatric rare diseases patients.

4.4. Statistical analyses, sample size 4.4.1. Statistical analysis Statistical analysis was planned in cooperation with the Institute of Medical Statistics Center for Medical Data Science, Medical University of Vienna.

First a t-test will be applied to test the primary objective: differences of participants' knowledge and well-being (Rare Disease Specific Self-Rating Scale) between the study time points T0 and T1, in the intervention group compared to the waitlist control group. For both groups, mean values and standard deviations will be reported. In case of a skewed distribution, a Wilcoxon test will be computed and median and interquartile range will be reported. The significance level will be set to 0.05. In case of missing values for study time point T1, for the primary analysis, only available cases will be considered. A sensitivity analysis will be performed to compare baseline data of patients with complete data and patients with missing data (descriptive statistics as only a small number of missing values is expected).

Tests for secondary endpoints: H2, H3 and H5 (difference in change in expert-rating scales, Quality of Life and mental health well-being, competences and mental health well-being) are analyzed in the same manner as the primary objective. To analyze the independent variables age, educational level and intellectual ability on the change in "Rare Disease Specific Self-Rating Scale", first univariate analyses of covariances (Ancova) will be computed and second a multiple Ancova will be performed with independent variables age, educational level and intellectual ability and group. For the secondary analyses, the significance level will be set to 0.05. No adjustment for multiplicity will be performed and p-values will be interpreted descriptively.

Descriptive statistics will be used to summarize baseline characteristics of recruited participants. Baseline characteristics will be presented in a table for the full enrolled sample. In order to test differences at baseline between the two groups with regard to theoretical and practical knowledge, as well as emotion t-tests for independent samples will be performed. The satisfaction with the Education & Care in RARE program for the intervention groups and for the applying experts (Patient Evaluation of the Education & Care in RARE program, at T1 and T2). Categorical variables will be presented in absolute frequencies and percentages. Continuous variables will be listed in means and standard deviations and will be presented in tables. Statistical analysis will be performed using SPSS 24 (IBM Corporation, Armonk, NY, USA).

4.4.2. Sample size calculation Sample size calculation was done for the primary study outcome "differences of participants' self-rating scales regarding knowledge about rare diseases and well-being (Rare Disease Specific Self-Rating Scale), before and after intervention with Education & Care in RARE". Sample size estimation was evaluated using R (Version 4.4.1, library pwr). We based the sample size calculation on parameters derived from some internal pilot data where we observed a standard deviation of 0.55 for the change between T0 and T1 (intervention group). However, as the study population will be very heterogenous (for example over 8.000 potential different rare diseases, high variability of knowledge on the underlying rare disease in the study population…) we consider more conservative estimates for the sample size calculation. These estimates should be considered as vague approximations. Thus, assuming that the standard deviation is equal for the intervention and the control group we performed several sample size calculations for standard deviations 0.55, 0.8, and 1 and several effect sizes (difference of differences) for a two-tailed t-test for independent groups (significance level 0.05 and power 0.8). The results can be found below. Based on this, sample size estimates indicate that we will be able to detect a difference of differences of 0.5 when the standard deviation of the difference in both groups is 0.8 with a sample size of 49 participants in each group and considering a dropout rate of 15%.

4.4.3. Methods of preventing bias Participants will be randomized using an online-randomization (https://www.meduniwien.ac.at/web/mitarbeiterinnen/it-hilfe-support/it4science/plattformen/randomizer/).

Patients will be randomized in blocks with random block lengths between 4 and 8 and stratified for center.¬¬ 4.4.5. Recruiting This prospective randomized controlled trial will be performed at several pediatric centers in Austria, which are involved in the diagnostics and care of pediatric rare diseases patients. In participating centers, during routine check-ups, patients who meet the inclusion and exclusion criteria, are invited to take part in the study.

Patients and their legal guardians are informed in detail about the study by the treating doctors or psychologist during a personal interview. There is written project information for children and adolescents of different age groups (age in years: 8-10, 11-14, 15-18, more than 18 years) and for parents/caregivers. If there are no more questions, written consent is obtained.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with a confirmed diagnosis of a rare disease with
* Age 5-20 years, corresponding to a developmental age of 5-18 years
* Existing medical care at a participating study center because of the rare disease
* Voluntary participation and informed consent
* Ability to complete the questionnaires
* Ability to actively participate the intervention (psychoeducation)

Exclusion Criteria:

* Moderate or severe cognitive impairment
* Simultaneous admission of the child / adolescent to a setting with high-frequency psychotherapeutic intervention (e.g. admission to psychosomatic medicine, child and adolescent psychiatry)
* No informed consent
* Language barrier of the child / adolescent
* Assumption that compliance is too low to attend all study appointments

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Rare Disease Specific Self-Rating Scale | IG: T0 (at inclusion), T1 (after intervention), T2 (3 to 6 months after T1); WLG: T0 (at inclusion), T1 (2-3 months after T0), T2 (after intervention), T3 (3 to 6 months after T2)
  Description:
  The Rare Disease Specific Self-Rating Scale is defined as primary outcome measurement of this study. The Rare Disease Specific Self-Rating Scale provides 10 items to assess rare disease specific knowledge and well-being in children and adolescents and uses a Six-Point Smiley Faces Likert Scale as a global subjective outcome scale for children assessment. For the primary hypothesis, a mean value of the 10 items is computed for each participant. The Rare Disease Specific Self-Rating Scale covers specific topics on Rare Diseases which are not covered by the generic research instruments of this study.
  Outcome Measurements:
  Knowledge about rare diseases; Well-being
  Items; Scale level:
  10 items; 6-Point Smiley Faces Likert Scale; sum total score 10-60;

SECONDARY OUTCOMES:
Rare Diseases Specific Expert-Rating Scale | IG: T0 (at inclusion), T1 (after intervention), T2 (3 to 6 months after T1); WLG: T0 (at inclusion), T1 (2-3 months after T0), T2 (after intervention), T3 (3 to 6 months after T2)
  Description:
  The Rare Disease Specific Expert-Rating Scale provides 12 items on participants' knowledge about rare diseases and on competences to cope with rare disease specific challenges and uses a Six-Point Smiley Faces Likert Scale as a global subjective outcome scale for expert assessment. For the analyses, a mean value of the 12 items is computed for each participant
  Outcome measurements:
  Knowledge about rare diseases, Competences to cope with rare disease specific challenges
  Items; Scales:
  12 items; 6-Point Smiley Faces Likert Scale; sum total score 12-72
SDQ Strengths and Difficulties Questionnaire self-report | IG: T0 (at inclusion), T1 (after intervention), T2 (3 to 6 months after T1); WLG: T0 (at inclusion), T1 (2-3 months after T0), T2 (after intervention), T3 (3 to 6 months after T2)
  Description:
  The SDQ Strengths and Difficulties Questionnaire (https://www.sdqinfo.org/a0.html) is a brief behavioral screening questionnaire in children and adolescents and provide 25 items on psychological attributes and includes a self-report version and a third-party survey version. There are two versions of the SDQ for two different age and development stages. A self-report version and a third-party survey version are offered for each age version of the SDQ. Norm values for different nationalities including German is available.
  Outcome Measurements:
  Mental health well-being - self-report
  Items; Scale level:
  25 items; 3-Point Likert Scale; sum total score 25-75
SDQ Strengths and Difficulties Questionnaire, third- party-report | IG: T0 (at inclusion), T2 (3 to 6 months after T1, T1 is defined as time point immideately after intervention); WLG: T0 (at inclusion), T1 (2-3 months after T0), T3 (3 to 6 months after T2, T2 is defined as time point immideately after intervention)
  Description:
  The SDQ Strengths and Difficulties Questionnaire (https://www.sdqinfo.org/a0.html) is a brief behavioral screening questionnaire in children and adolescents and provide 25 items on psychological attributes and includes a self-report version and a third-party survey version. There are two versions of the SDQ for two different age and development stages. A self-report version and a third-party survey version are offered for each age version of the SDQ. Norm values for different nationalities including German is available.
  Outcome Measurements:
  Mental health well-being - third-party-report
  Items; Scale level:
  25 items; 3-Point Likert Scale; sum total score 25-75
KINDL self-report | IG: T0 (at inclusion), T1 (after intervention), T2 (3 to 6 months after T1); WLG: T0 (at inclusion), T1 (2-3 months after T0), T2 (after intervention), T3 (3 to 6 months after T2)
  Description: The KINDL (https://www.kindl.org/english/) is a standardized questionnaire for the assessment of quality of life in children and adolescents and provides 24 items. The KINDL thus is a short, methodologically suitable, psychometrically sound and flexible measure of Health-Related Quality of Life in children and adolescents. There are three versions of the KINDL for different age and development stages. A self-report version and a third-party survey version are offered for each age version of the KINDL. Norm values are given based on representative German data from the German National Health Interview and Examination Survey for Children and Adolescents (KiGGS). The KiGGS study is a broad survey realized by the German-Robert-Koch-Institute.
  Outcome Measurements:
  Quality of life - self-report
  Items; Scale level:
  24 items; 3-Point Likert Scale; sum total score 24-72
KINDL third-party-report | IG: T0 (at inclusion), T2 (3 to 6 months after T1, T1 is defined as time point immideately after intervention); WLG: T0 (at inclusion), T1 (2-3 months after T0), T3 (3 to 6 months after T2, T2is defined as time point immideately after intervention)
  Description: The KINDL (https://www.kindl.org/english/) is a standardized questionnaire for the assessment of quality of life in children and adolescents and provides 24 items. The KINDL thus is a short, methodologically suitable, psychometrically sound and flexible measure of Health-Related Quality of Life in children and adolescents. There are three versions of the KINDL for different age and development stages. A self-report version and a third-party survey version are offered for each age version of the KINDL. Norm values are given based on representative German data from the German National Health Interview and Examination Survey for Children and Adolescents (KiGGS). The KiGGS study is a broad survey realized by the German-Robert-Koch-Institute.
  Outcome Measurements:
  Quality of life - third-party-report
  Items; Scale level:
  24 items; 3-Point Likert Scale; sum total score 24-72
Patients' evaluation of the Education & Care in RARE Program | IG: T1 (after intervention); WLG T2 (after intervention)
  Description:
  The Patient Evaluation of the Education & Care in RARE program provides 3 items to assess attractiveness, helpfulness, and recommendability of the program and uses a Six-Point Smiley Faces Likert Scale as a global subjective outcome scale for expert assessment.
  Outcome Measurements:
  Program evaluation by patients: attractiveness; helpfulness; recommendability;
  Items; Scale level:
  3 items, 6-Point Smiley Faces Likert Scale; descriptive
Expert Evaluation of the Education & Care in RARE program | IG: T1 (after intervention); WLG T2 (after intervention)
  Description:
  The Expert Evaluation of the Education & Care in RARE program provides 10 items to assess the degree of achievement of specific psychosocial therapeutic goals of the program and uses a Three-Point Likert Scale as a global subjective outcome scale for expert assessment. As no guidelines for the psychosocial care in rare diseases exists - the defined items are adapted according to S3 Guideline Psychosocial care in pediatric oncology and hematology and include following psychosocial goals: Gaining information; Promoting the ability to act and co-operation; Strengthening the individual resources competences and autonomy; Promotion of coping strategies; Strengthening self-esteem; Supporting open communication; Promoting verbal and non-verbal expression; Promotion of understanding of the illness; Promoting the best possible health-related quality of life and mental health; Reduction of fear, powerlessness; Items: Scale: 10 items, 3-Point Likert Scale; descriptive

OTHER OUTCOMES:
Documentation of the program | IG: T2 (at last follow up, 3 to 6 months after T1, T1 is defined as time point immediately after intervention); WLG: T3 (last follow up, 3 to 6 months after T1, T1 is defined as time point immediately after intervention))
  Documentation of the program provides number of sessions and levels of the Education & Care in RARE program in each participant.
  Items; Scales:
  2 items, descriptive
Medical Data | IG: after inclusion WLG: after inclusion
  Medical Data asses medical data of study participants including Rare disease diagnosis Secondary conditions Developmental age Visibility of a rare disease Type of visibility of a rare disease Type of diagnostic confirmation Life-threatening rare disease Age at rare disease diagnosis Time of diagnostic odyssey Existence of an emergency card or a rare disease card
  Items; Scales:
  10 items, descriptive
Demographic Data | IG: after inclusion WLG: after inclusion
  Participants sociodemographic data including Patient's age, sex, school form, language skills, mother language, multilingualism; Parents' education and language skills;
  Items; Scales:
  8 items, descriptive

CONTACTS AND LOCATIONS:
Locations (7):
- Austria (7):
  - Medical University of Graz, Graz, Austria
  - Medical University of Innsbruck, Innsbruck, Austria
  - The Faculty of Medicine JKU Linz, Linz, Austria
  - SALK PMU, Salzburg, Austria
  - WIGEV Klinikum Favoriten, Vienna, Austria
  - Ordensklinikum Linz, Linz
  - Medical University of Vienna, Vienna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Temizsoy H, Ozlu-Erkilic Z, Ohmann S, Sackl-Pammer P, Popow C, Akkaya-Kalayci T. Influence of Psychopharmacotherapy on the Quality of Life of Children with Attention-Deficit/Hyperactivity Disorder. J Child Adolesc Psychopharmacol. 2019 Aug;29(6):419-425. doi: 10.1089/cap.2018.0131. Epub 2019 Mar 29. PMID 30925091
- [Background] Sackl-Pammer P, Ozlu-Erkilic Z, Jahn R, Karwautz A, Pollak E, Ohmann S, Akkaya-Kalayci T. Somatic complaints in children and adolescents with social anxiety disorder. Neuropsychiatr. 2018 Dec;32(4):187-195. doi: 10.1007/s40211-018-0288-8. Epub 2018 Sep 14. PMID 30218392
- [Background] Sackl-Pammer P, Jahn R, Ozlu-Erkilic Z, Pollak E, Ohmann S, Schwarzenberg J, Plener P, Akkaya-Kalayci T. Social anxiety disorder and emotion regulation problems in adolescents. Child Adolesc Psychiatry Ment Health. 2019 Sep 30;13:37. doi: 10.1186/s13034-019-0297-9. eCollection 2019. PMID 31583014
- [Background] Ohmann S, Popow C, Wurzer M, Karwautz A, Sackl-Pammer P, Schuch B. Emotional aspects of anorexia nervosa: results of prospective naturalistic cognitive behavioral group therapy. Neuropsychiatr. 2013;27(3):119-28. doi: 10.1007/s40211-013-0065-7. Epub 2013 Jun 18. PMID 23775391
- [Background] Vodopiutz J, Schmook MT, Konstantopoulou V, Plecko B, Greber-Platzer S, Creus M, Seidl R, Janecke AR. MED20 mutation associated with infantile basal ganglia degeneration and brain atrophy. Eur J Pediatr. 2015 Jan;174(1):113-8. doi: 10.1007/s00431-014-2463-7. Epub 2014 Dec 3. PMID 25446406
- [Background] Breu M, Hafele C, Trimmel-Schwahofer P, Schmidt WM, Laconne F, Vodopiutz J, Male C, Dressler A. The relation of etiology based on the 2017 ILAE classification to the effectiveness of the ketogenic diet in drug-resistant epilepsy in childhood. Epilepsia. 2021 Nov;62(11):2814-2825. doi: 10.1111/epi.17052. Epub 2021 Aug 28. PMID 34453316
- [Background] Ritter M, Vodopiutz J, Lechner S, Moser E, Schmidt-Erfurth UM, Janecke AR. Coexistence of KCNV2 associated cone dystrophy with supernormal rod electroretinogram and MFRP related oculopathy in a Turkish family. Br J Ophthalmol. 2013 Feb;97(2):169-73. doi: 10.1136/bjophthalmol-2012-302355. Epub 2012 Nov 10. PMID 23143909
- [Background] Siegert S, Mindler GT, Brucke C, Kranzl A, Patsch J, Ritter M, Janecke AR, Vodopiutz J. Expanding the Phenotype of the FAM149B1-Related Ciliopathy and Identification of Three Neurogenetic Disorders in a Single Family. Genes (Basel). 2021 Oct 20;12(11):1648. doi: 10.3390/genes12111648. PMID 34828254
- [Background] Walleczek NK, Forster K, Seyr M, Kadrnoska N, Kolar J, Wasinger-Brandweiner V, Vodopiutz J. Rare skeletal disorders: a multidisciplinary postnatal approach to diagnosis and management. Wien Med Wochenschr. 2021 Apr;171(5-6):94-101. doi: 10.1007/s10354-021-00820-2. Epub 2021 Mar 10. PMID 33689085
- [Background] Vodopiutz J, Zoller H, Fenwick AL, Arnhold R, Schmid M, Prayer D, Muller T, Repa A, Pollak A, Aufricht C, Wilkie AO, Janecke AR. Homozygous SALL1 mutation causes a novel multiple congenital anomaly-mental retardation syndrome. J Pediatr. 2013 Mar;162(3):612-7. doi: 10.1016/j.jpeds.2012.08.042. Epub 2012 Oct 12. PMID 23069192
- [Background] Muller T, Mizumoto S, Suresh I, Komatsu Y, Vodopiutz J, Dundar M, Straub V, Lingenhel A, Melmer A, Lechner S, Zschocke J, Sugahara K, Janecke AR. Loss of dermatan sulfate epimerase (DSE) function results in musculocontractural Ehlers-Danlos syndrome. Hum Mol Genet. 2013 Sep 15;22(18):3761-72. doi: 10.1093/hmg/ddt227. Epub 2013 May 23. PMID 23704329
- [Background] McInerney-Leo AM, Harris JE, Leo PJ, Marshall MS, Gardiner B, Kinning E, Leong HY, McKenzie F, Ong WP, Vodopiutz J, Wicking C, Brown MA, Zankl A, Duncan EL. Whole exome sequencing is an efficient, sensitive and specific method for determining the genetic cause of short-rib thoracic dystrophies. Clin Genet. 2015 Dec;88(6):550-7. doi: 10.1111/cge.12550. Epub 2015 Feb 17. PMID 25492405
- [Background] Jansen EJ, Timal S, Ryan M, Ashikov A, van Scherpenzeel M, Graham LA, Mandel H, Hoischen A, Iancu TC, Raymond K, Steenbergen G, Gilissen C, Huijben K, van Bakel NH, Maeda Y, Rodenburg RJ, Adamowicz M, Crushell E, Koenen H, Adams D, Vodopiutz J, Greber-Platzer S, Muller T, Dueckers G, Morava E, Sykut-Cegielska J, Martens GJ, Wevers RA, Niehues T, Huynen MA, Veltman JA, Stevens TH, Lefeber DJ. ATP6AP1 deficiency causes an immunodeficiency with hepatopathy, cognitive impairment and abnormal protein glycosylation. Nat Commun. 2016 May 27;7:11600. doi: 10.1038/ncomms11600. PMID 27231034
- [Background] Holt-Danborg L, Vodopiutz J, Nonboe AW, De Laffolie J, Skovbjerg S, Wolters VM, Muller T, Hetzer B, Querfurt A, Zimmer KP, Jensen JK, Entenmann A, Heinz-Erian P, Vogel LK, Janecke AR. SPINT2 (HAI-2) missense variants identified in congenital sodium diarrhea/tufting enteropathy affect the ability of HAI-2 to inhibit prostasin but not matriptase. Hum Mol Genet. 2019 Mar 1;28(5):828-841. doi: 10.1093/hmg/ddy394. PMID 30445423
- [Background] Dundar M, Muller T, Zhang Q, Pan J, Steinmann B, Vodopiutz J, Gruber R, Sonoda T, Krabichler B, Utermann G, Baenziger JU, Zhang L, Janecke AR. Loss of dermatan-4-sulfotransferase 1 function results in adducted thumb-clubfoot syndrome. Am J Hum Genet. 2009 Dec;85(6):873-82. doi: 10.1016/j.ajhg.2009.11.010. PMID 20004762
- [Background] Diets IJ, van der Donk R, Baltrunaite K, Waanders E, Reijnders MRF, Dingemans AJM, Pfundt R, Vulto-van Silfhout AT, Wiel L, Gilissen C, Thevenon J, Perrin L, Afenjar A, Nava C, Keren B, Bartz S, Peri B, Beunders G, Verbeek N, van Gassen K, Thiffault I, Cadieux-Dion M, Huerta-Saenz L, Wagner M, Konstantopoulou V, Vodopiutz J, Griese M, Boel A, Callewaert B, Brunner HG, Kleefstra T, Hoogerbrugge N, de Vries BBA, Hwa V, Dauber A, Hehir-Kwa JY, Kuiper RP, Jongmans MCJ. De Novo and Inherited Pathogenic Variants in KDM3B Cause Intellectual Disability, Short Stature, and Facial Dysmorphism. Am J Hum Genet. 2019 Apr 4;104(4):758-766. doi: 10.1016/j.ajhg.2019.02.023. Epub 2019 Mar 28. PMID 30929739
- [Background] Vodopiutz J, Seidl R, Prayer D, Khan MI, Mayr JA, Streubel B, Steiss JO, Hahn A, Csaicsich D, Castro C, Assoum M, Muller T, Wieczorek D, Mancini GM, Sadowski CE, Levy N, Megarbane A, Godbole K, Schanze D, Hildebrandt F, Delague V, Janecke AR, Zenker M. WDR73 Mutations Cause Infantile Neurodegeneration and Variable Glomerular Kidney Disease. Hum Mutat. 2015 Nov;36(11):1021-8. doi: 10.1002/humu.22828. Epub 2015 Aug 6. PMID 26123727
- [Background] Vodopiutz J, Mizumoto S, Lausch E, Rossi A, Unger S, Janocha N, Costantini R, Seidl R, Greber-Platzer S, Yamada S, Muller T, Jilma B, Ganger R, Superti-Furga A, Ikegawa S, Sugahara K, Janecke AR. Chondroitin Sulfate N-acetylgalactosaminyltransferase-1 (CSGalNAcT-1) Deficiency Results in a Mild Skeletal Dysplasia and Joint Laxity. Hum Mutat. 2017 Jan;38(1):34-38. doi: 10.1002/humu.23070. Epub 2016 Sep 22. PMID 27599773
- [Background] Braunholz D, Obieglo C, Parenti I, Pozojevic J, Eckhold J, Reiz B, Braenne I, Wendt KS, Watrin E, Vodopiutz J, Rieder H, Gillessen-Kaesbach G, Kaiser FJ. Hidden mutations in Cornelia de Lange syndrome limitations of sanger sequencing in molecular diagnostics. Hum Mutat. 2015 Jan;36(1):26-9. doi: 10.1002/humu.22685. Epub 2014 Dec 2. PMID 25196272
- [Background] Waich S, Janecke AR, Parson W, Greber-Platzer S, Muller T, Huber LA, Valovka T, Vodopiutz J. Novel PCNT variants in MOPDII with attenuated growth restriction and pachygyria. Clin Genet. 2020 Sep;98(3):282-287. doi: 10.1111/cge.13797. Epub 2020 Jul 7. PMID 32557621
- [Background] Waich S, Roscher A, Brunner-Krainz M, Cortina G, Kostl G, Feichtinger RG, Entenmann A, Muller T, Knisely AS, Mayr JA, Janecke AR, Vodopiutz J. Severe Deoxyguanosine Kinase Deficiency in Austria: A 6-Patient Series. J Pediatr Gastroenterol Nutr. 2019 Jan;68(1):e1-e6. doi: 10.1097/MPG.0000000000002149. PMID 30589726
- [Background] Witt S, Kristensen K, Wiegand-Grefe S, Boettcher J, Bloemeke J, Wingartz C, Bullinger M, Quitmann J; und die CARE-FAM-NET Studiengruppe. Rare pediatric diseases and pathways to psychosocial care: a qualitative interview study with professional experts working with affected families in Germany. Orphanet J Rare Dis. 2021 Nov 27;16(1):497. doi: 10.1186/s13023-021-02127-2. PMID 34838091
- [Background] Baldovino S, Moliner AM, Taruscio D, Daina E, Roccatello D. Rare Diseases in Europe: from a Wide to a Local Perspective. Isr Med Assoc J. 2016 Jun;18(6):359-63. PMID 27468531
- See also: Related Info — https://www.orpha.net/en/other-information/about-rare-diseases
- See also: Related Info — https://ccp.meduniwien.ac.at/patienteninfo/informationen-fuer-kinder-und-jugendliche/cartoon-ein-psychoedukatives-schulungsprogramm/
- See also: Related Info — https://www.youtube.com/watch?v=R3fr-q-6JIw
- See also: Related Info — https://kinder-jugendheilkunde.meduniwien.ac.at/informationen-fuer-patientinnen/education-care-in-rare/